CLINICAL TRIAL: NCT02488070
Title: 68Ga-PSMA PET/CT or PET/MRI in the Evaluation of Patients With Prostate Cancer: A Feasibility Study
Brief Title: 68Ga-PSMA PET/CT or PET/MRI in Evaluating Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-32985; NCI-2015-01067 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PROS0068 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (68Ga-PSMA PET/CT or PET/MRI) (Experimental): Patients receive gallium Ga 68-labeled PSMA ligand Glu-urea-Lys(Ahx) IV and then undergo PET/CT or PET/MRI approximately 45-60 minutes later.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-labeled PSMA Ligand Glu-urea-Lys(Ahx); Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Part of PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Drug: Gallium Ga 68-labeled PSMA Ligand Glu-urea-Lys(Ahx) — Intravenously-administered (IV) radioisotope
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-HBED-CC-PSMA; ProstaMedix
Procedure: Magnetic Resonance Imaging — Part of PET/MRI scan
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Part of PET/CT and/or PET/MRI scans
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies gallium-68 (68Ga)-prostate specific membrane antigen (PSMA) (gallium Ga 68-labeled PSMA ligand Glu-urea-Lys[Ahx]) positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI) in identifying prostate cancer that may have returned after a period of improvement (biochemical recurrence). 68Ga-PSMA is a radiopharmaceutical that localizes to a specific prostate cancer receptor, which can then be imaged by the PET/CT or PET/MRI scanner.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Evaluate the feasibility and biodistribution of 68Ga-PSMA.

OUTLINE:

Patients are injected with 5 mCi of Ga68 PSMA intravenously (IV) and then undergo PET/CT or PET/MRI approximately 45 to 60 minutes later.

After completion of study, patients are followed up at 24 hours and 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Known diagnosis of prostate cancer
* Patient has suspected recurrence based on biochemical data (prostate specific antigen [PSA] > 2 ng/mL)
* Able to remain still for duration of each imaging procedure (about one hour)

Exclusion Criteria:

* Unable to provide informed consent
* Inability to lie still for the entire imaging time
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afshar-Oromieh A, Malcher A, Eder M, Eisenhut M, Linhart HG, Hadaschik BA, Holland-Letz T, Giesel FL, Kratochwil C, Haufe S, Haberkorn U, Zechmann CM. PET imaging with a [68Ga]gallium-labelled PSMA ligand for the diagnosis of prostate cancer: biodistribution in humans and first evaluation of tumour lesions. Eur J Nucl Med Mol Imaging. 2013 Apr;40(4):486-95. doi: 10.1007/s00259-012-2298-2. Epub 2012 Nov 24. PMID 23179945
- [Result] Minamimoto R, Hancock S, Schneider B, Chin FT, Jamali M, Loening A, Vasanawala S, Gambhir SS, Iagaru A. Pilot Comparison of (6)(8)Ga-RM2 PET and (6)(8)Ga-PSMA-11 PET in Patients with Biochemically Recurrent Prostate Cancer. J Nucl Med. 2016 Apr;57(4):557-62. doi: 10.2967/jnumed.115.168393. Epub 2015 Dec 10. PMID 26659347

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (68Ga-PSMA PET/CT or PET/MRI): Patients receive gallium Ga 68-labeled PSMA ligand Glu-urea-Lys(Ahx) IV and then undergo PET/CT or PET/MRI approximately 45-60 minutes later.
  Computed Tomography: Undergo PET/CT
  Gallium Ga 68-labeled PSMA Ligand Glu-urea-Lys(Ahx): Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Magnetic Resonance Imaging: Undergo PET/MRI
  Positron Emission Tomography: Undergo PET/CT
  Positron Emission Tomography: Undergo PET/MRI
Period: Overall Study
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Average SUVmax of Ga68 PSMA Uptake Outside the Expected Normal Biodistribution
Description: The biodistribution (ie, the location(s) of physiologic radiopharmaceutical uptake within the body) of Ga68 PSMA will be evaluated using PET/CT or PET/MRI. Biodistribution will be measured by drawing regions of interest (ROI) around areas with visually appreciable increased focal uptake over background (mediastinal blood pool) and calculating a standardized uptake value maximum (SUVmax), which is a semi-quantitative measurement of the maximum value of radiopharmaceutical uptake within the ROI.
Time Frame: an estimated average of 1 hour
Population: 45 areas of high Ga68 PSMA focal uptake outside the normal biodistribution were used to calculate the average SUVmax. The mediastinal blood pool was used to determine average background.
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
Number analyzed (Participants) | 10
SUVmax | 12.4 (7.1)

2. Primary Outcome: Average SUVmean of Ga68 PSMA Uptake Outside the Expected Normal Biodistribution
Description: The biodistribution (ie, the location(s) of physiologic radiopharmaceutical uptake within the body) of Ga68 PSMA will be evaluated using PET/CT or PET/MRI. Biodistribution will be measured by drawing regions of interest (ROI) around areas with visually appreciable increased focal uptake over background (mediastinal blood pool) and calculating a SUVmean which is a semi-quantitative measurement of the average value of radiopharmaceutical uptake within the ROI.
Time Frame: an estimated average of 1 hour
Population: 45 areas of high Ga68 PSMA focal uptake outside the normal biodistribution were used to calculate the average SUVmean. The mediastinal blood pool was used to determine average background.
Measure: Mean (Standard Deviation); unit: SUVmean
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
Number analyzed (Participants) | 10
SUVmean | 7.1 (4.0)

3. Primary Outcome: Average SUVmax Focal Uptake of Ga68 PSMA (F/N Ratio)
Description: Focal uptake will be measured by drawing regions-of-interest (ROI) around areas with visually appreciable increased focal uptake over background (mediastinal blood pool) and calculating a SUVmax (a semi-quantitative measurement of the maximum value of radiopharmaceutical uptake within the ROI). The result will be expressed as the F/N ratio, ie, SUVmax of focal uptake divided by SUVmax of background.
Time Frame: an estimated average of 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: F/N ratio
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
Number analyzed (Participants) | 10
F/N ratio | 10.4 (9.3)

4. Primary Outcome: Average SUVmean Focal Uptake of Ga68 PSMA (F/N Ratio)
Description: Focal uptake will be measured by drawing regions-of-interest (ROI) around areas with visually appreciable increased focal uptake over background (mediastinal blood pool) and calculating a SUVmean (a semi-quantitative measurement of the average value of radiopharmaceutical uptake within the ROI). The result will be expressed as the F/N ratio, ie, SUVmax of focal uptake divided by SUVmax of background.
Time Frame: an estimated average of 1 hour
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: F/N ratio
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
Number analyzed (Participants) | 10
F/N ratio | 9.2 (7.3)

5. Secondary Outcome: Feasibility of Ga-68 PSMA PET/CT or PET/MRI Scan
Description: Feasibility of Ga68 PSMA PET/CT or PET/MRI is expressed as the number of subjects for whom the scan was successfully completed.
Time Frame: an estimated average of 2 hours
Population: The population analyzed included all participants receiving Ga-68 PSMA PET/CT or PET/MRI scan.
Measure: Number; unit: participants
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Arm/Group | Diagnostic (68Ga-PSMA PET/CT or PET/MRI)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
lack of correlation with pathology results for all patients; limited patient enrollment (pilot study)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes